CLINICAL TRIAL: NCT01731483
Title: Coagulation and Fibrinolysis as Virulence Factors for Invasive Staphylococcus Aureus and Streptococcus Infections.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Peter Verhamme, Prof. Verhamme, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: M-1
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Infective Endocarditis; Necrotizing Fasciitis
Keywords: virulence factors
MeSH Terms: conditions — Endocarditis; Fasciitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue specimens from endocarditis lesions and necrotizing fasciitis
Oversight: Data Monitoring Committee: No

SUMMARY:
the aim of this study is to investigate the role of staphylokinase, streptokinase and MMP activation in invasive staphylococcal and streptococcal infections.

ELIGIBILITY:
Inclusion Criteria:

* all patients that undergo surgical treatment for invasive streptococcal or staphylococcal infections, including acute infective endocarditis and necrotizing fasciitis, from the UZ Leuven University Hospital

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Material will be collected from all patients that undergo surgical treatment for invasive streptococcal or staphylococcal infections, including acute infective endocarditis and necrotizing fasciitis, from the UZ Leuven University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2012-07; Primary Completion 2020-03 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
proteolytic activity | 1 day (on date of surgery (tissue sample))

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verhamme, MD,PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven University Hospital, Leuven, Belgium